CLINICAL TRIAL: NCT06484335
Title: RV630 - Approach to Control HIV With Immune Enhancement and Vaccination (ACHIEV): Safety and Efficacy of Broadly Neutralizing Antibodies Combined With Therapeutic Vaccination for the Induction of HIV Remission
Brief Title: RV630 - Approach to Control HIV With Immune Enhancement and Vaccination (ACHIEV
Acronym: ACHIEV
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: US Military HIV Research Program (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RV 630/ACHIEV
Record Dates: First submitted 2024-05-31; First posted 2024-07-03 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: HIV Infections; PLWH; ART; Acute HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The participants, clinical staff, laboratory staff, Principal Investigator (PI) and the Sponsor will be blinded to vaccine/placebo allocation for Groups 1 and 2. The pharmacist with primary responsibility for vaccine dispensing will not be blinded to the treatment and maintains the randomization code and completes assignments of participants according to the randomization allocation.
  The contents of the syringes containing vaccine IP will be obscured and not discernable to the participant or study staff in the vaccination room. All analyses conducted prior to the completion of the study will be performed by an unblinded statistician, and results will only be presented in aggregate to protect the participant-level blind. See Section 6.4 below for unblinding procedures.
  Group 3 will be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Active Arm (Active Comparator): Active Arm (Group 1) will have 20 participants. For the primary objectives and endpoints, this study will enroll participants of the RV 254/WRAIR #1494 study, who are PLWH aged 18 - 60 years, initiated ART during Fiebig I-V AHI, are virologically suppressed (HIV-1 RNA < 50 copies/mL for ≥ 48 weeks) on uninterrupted ART, and who meet study inclusion criteria into Groups 1 and 2. For Active Arm: Group 1 will receive:
  i. VRC07-523LS and PGDM1400LS at Step 2, Week 0 ii. ART starting at Step 2, Week 1 iii. ChAdOx1.tHIVconsv1 and ChAdOx1.HIVconsv62 vaccination at Step 2, Week 4 iv. MVA.tHIVconsv4 and A244d11 gp120/ALFQ vaccination at Step 2, Weeks 12 and 20
  Interventions: Biological: VRC07-523LS; Biological: PGDM1400LS; Biological: ChAdOx1.tHIVconsv1; Biological: ChAdOx1.HIVconsv62; Biological: MVA.tHIVconsv4; Biological: A244d11 gp120; Biological: ALFQ
- Comparator Arm (Placebo Comparator): Comparator Arm (Group 2) will have 20 participants. For the primary objectives and endpoints, this study will enroll participants of the RV 254/WRAIR #1494 study, who are PLWH aged 18 - 60 years, initiated ART during Fiebig I-V AHI, are virologically suppressed (HIV-1 RNA < 50 copies/mL for ≥ 48 weeks) on uninterrupted ART, and who meet study inclusion criteria into Groups 1 and 2. For Comparator Arm - Group 2 will receive:
  i. VRC07-523LS and PGDM1400LS at Step 2, Week 0 ii. ART starting at Step 2, Week 1 iii. Placebo vaccination at Step 2, Weeks 4, 12 and 20
  Interventions: Biological: VRC07-523LS; Biological: PGDM1400LS; Other: Placebo
- Exploratory Arm (Other): Exploratory Arm (Group 3) will have 8 participants. This study will also enroll an Exploratory arm of newly enrolled participants of the RV 254/ WRAIR #1494 study, who are PLWH aged 18 - 60 years, diagnosed during Fiebig I-V AHI, have not yet initiated ART, and meet all study inclusion criteria into Group 3.
  For the Exploratory Arm - Group 3 will receive:
  iv. VRC07-523LS and PGDM1400LS at Step 2, Week 0 v. ART starting at Step 2, Week 0 vi. ChAdOx1.tHIVconsv1 and ChAdOx1.HIVconsv62 vaccination at Step 2, Week 12 vii. MVA.tHIVconsv4 and A244d11 gp120/ALFQ vaccination at Step 2, Weeks 20 and 28
  Interventions: Biological: VRC07-523LS; Biological: PGDM1400LS; Biological: ChAdOx1.tHIVconsv1; Biological: ChAdOx1.HIVconsv62; Biological: MVA.tHIVconsv4; Biological: A244d11 gp120; Biological: ALFQ

INTERVENTIONS:
Biological: VRC07-523LS — VRC07-523LS (VRC-HIVMAB075-00-AB) is a recombinant human immunoglobulin G1 (IgG1) broadly neutralizing monoclonal antibody (bNAb) directed against the HIV-1 CD4 binding site
Biological: PGDM1400LS — PGDM1400LS is a recombinant human IgG1 bNAb targeted against the HIV-1 V2 apex epitope region.
Biological: ChAdOx1.tHIVconsv1 — ChAdOx1.tHIVconsv1 is a replication-deficient virus expressing six conserved sub-protein regions of Gag and Pol (regions 1-6) of HIV-1 as one chimeric protein designated HIVconsv1.
  Arms: Active Arm; Exploratory Arm
Biological: ChAdOx1.HIVconsv62 — ChAdOx1.HIVconsv62 is a replication-deficient virus expressing six conserved sub-protein regions of Gag and Pol (regions 1-6) of HIV-1 as one chimeric protein designated HIVconsv62.
  Arms: Active Arm; Exploratory Arm
Biological: MVA.tHIVconsv4 — MVA.tHIVconsv4 is a recombinant, non-replicating Modified Vaccinia Ankara (MVA) virus expressing six conserved sub-protein regions of Gag and Pol (regions 1-6) of HIV-1 as one chimeric protein designated tHIVconsv4.
  Arms: Active Arm; Exploratory Arm
Biological: A244d11 gp120 — A244d11 gp120, consists of the gp120 envelope glycoprotein HIV-1 subtype CRF_01AE A244 derived from the CM244 CRF_01AE strain, with an 11 amino N-terminal deletion. It is a modification of the A244 rgp120 immunogen from the AIDSVAX®B/E vaccine.
  Arms: Active Arm; Exploratory Arm
Biological: ALFQ — ALFQ (Army Liposome Formulation, ALF) is a liposomal adjuvant containing a synthetic
  Arms: Active Arm; Exploratory Arm
Other: Placebo — Normal saline (0.9% sodium chloride for injection) will be used as a placebo.
  Arms: Comparator Arm

SUMMARY:
This is a phase I, randomized, double-blind, placebo-controlled clinical trial to investigate the safety of VRC07-523LS and PGDM1400LS in combination with ChAdOx1.tHIVconsv1, ChAdOx1.HIVconsv62 prime, MVA.tHIVconsv4 and A244d11gp120/ALFQ vaccination, and the impact on viral load setpoint during analytic treatment interruption (ATI) in people living with human immunodeficiency virus-1 (HIV-1, PLWH) who have initiated or will initiate antiretroviral therapy (ART) during acute HIV-1 infection (AHI).

DETAILED DESCRIPTION:
This is a phase I, randomized, double-blinded, placebo-controlled clinical trial to investigate the safety of VRC07-523LS and PGDM1400LS in combination with ChAdOx1.tHIVconsv1, ChAdOx1.tHIVconsv62, MVA.tHIVconsv4 and A244d11 gp120/ALFQ vaccination, and the impact on viral load setpoint during ATI in PLWH who initiated ART during AHI.

To evaluate the primary objectives, the study will enroll up to 40 adults already enrolled in the RV 254/WRAIR #1494 study who initiated ART during Fiebig I-V acute HIV-1 infection, with plasma HIV-1 RNA < 50 copies/mL for ≥ 48 weeks, CD4 T-cell counts ≥ 400 cells/mm3, viruses susceptible to VRC07-523LS and/or PGDM1400LS, and the absence of known protective HLA allele (Groups 1 and 2).

Participants currently on ART who meet study entry criteria will be randomized (Section 6.2) in a 1:1 allocation to the Active (Group 1) or Comparator (Group 2) Arms prior to entering Step 1.

To evaluate exploratory objectives, the study will also enroll up to 8 adults who are newly enrolled in the RV 254/WRAIR #1494 study, diagnosed during Fiebig I-V AHI, and have not yet initiated ART (Group 3).

ELIGIBILITY:
Inclusion/Exclusion Step 1 Inclusion Criteria (Groups 1 and 2 only)

Participants are eligible to be included in the protocol Step 1 only if all of the following criteria are met:

1. Thai National
2. Age ≥18 and ≤60 years of age
3. Can read and write Thai
4. Able and willing to provide written informed consent
5. Confirmed HIV-1 infection (nucleic acid testing [NAT] and/or HIV-1 serology positive with confirmatory quantitative HIV-1 viral load) and started ART during acute infection
6. Uninterrupted treatment with ART (no interruption of ART for ≥7 consecutive days or longer) since ART initiation, for ≥ 48 weeks.
7. Currently on integrase inhibitor-based ART regimen (excluding long-acting injectable regimens) and no recent (≤8 weeks prior to screening) changes to ART regimen.

   a. There must be at least one documented plasma HIV-1 RNA <50 cps/mL after the last ART change prior to screening
8. Must be medically stable as confirmed by medical history, physical examination, vital signs, and clinical laboratory tests performed at screening, and as per the Investigator's discretion.

   a. If the results of the screening laboratory panel are outside the normal reference ranges, the participant may be included only if the Investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study after discussion with the Sponsor's Representative.
9. The following laboratory values at screening:

   1. CD4 T-cell count ≥400 cells/mm3
   2. Absolute neutrophil count (ANC) ˃1,000/mm3
   3. Hemoglobin >11.5 g/dL
   4. Platelet count ˃150,000/mm3
   5. Estimated glomerular filtration rate (eGFR) ≥60 mL/min/1.73m2 using the re-expressed MDRD equation with Thai racial factor or the CKD-EPI Cystatin C equation.
   6. Aspartate aminotransferase (AST) (SGOT), alanine aminotransferase (ALT) (SGPT), alkaline phosphatase (AP), and total bilirubin ≤1.5 x the upper limit of normal (ULN)
   7. Hepatitis C virus (HCV) antibody negative or HCV RNA negative.
10. HIV-1 RNA <50 copies/ml for ≥48 weeks at screening.

    1. No history of virologic failure. Virologic failure is defined as having two consecutive HIV-1 RNA >1000 copies/mL at any time after achieving HIV-1 RNA <50 copies/mL
    2. A single viral load measurement ≥50 but <1000 copies/mL, at any time from achieving HIV-1 RNA <50 copies/mL to > 48 weeks from screening, is allowed provided that it is bracketed by viral loads <50 copies/mL
    3. A single viral load measurements ≥50 but <200 copies/mL, within 48 weeks of screening is allowed provided that each is bracketed by viral loads <50 copies/mL prior to screening.
11. Sensitivity test demonstrating the lack of detection of resistant viruses to VRC07-523LS or PGDM1400LS.
12. For persons of childbearing potential, negative pregnancy test at the screening visit.
13. Persons of childbearing potential must agree to not become pregnant and use two methods of contraception if engaging in sexual activity that could lead to pregnancy.
14. Participants engaging in sexual activity that could lead to pregnancy in the partner and who are of reproductive potential must agree to use a condom to avoid pregnancy in a spouse or partner of childbearing potential and to avoid transmitting HIV to an uninfected partner. A condom must be used from the time of screening until the end of the study or until viral suppression in Step 4, whichever occurs first.
15. Willingness to abstain from sexual intercourse, or use a condom, or partner(s) using preexposure prophylaxis consistently during ATI and until plasma HIV-1 RNA is less than limit of detection after ART restart with all partners that are HIV-uninfected or serostatus unknown.
16. Passes Test of Understanding (Protocol Section 8.4)
17. Willing to interrupt and restart ART according to study schedule
18. Willing to participate and adhere to the prohibitions and restrictions specified in this protocol for the duration of the study visits and follow up. Step 1 Exclusion Criteria (Groups 1 and 2 only)

Participants who meet any of the following criteria will be excluded from the study:

1. Weight <50 kg or > 115 kg
2. Presence of HLA B*57:01 allele associated with viral control.
3. Anyone with contraindication to intramuscular injections, placement of intravenous lines, and blood draws
4. Acute or serious illness requiring systemic treatment and/or hospitalization within 90 days prior to entry.
5. Any clinically significant acute or chronic medical condition, that in the opinion of the investigator would preclude participation including cardiovascular, pulmonary, hepatic, renal, gastrointestinal, genitourinary, hematological, coagulation, immunological disorders, that in the opinion of the investigator would preclude participation (e.g., history of seizure disorders, cardiovascular disease, bleeding/clotting disorder, autoimmune disease, malignancy, poorly controlled asthma, active tuberculosis or other systemic infections, etc.).
6. Active or chronic hepatitis B virus infection (detectable HBsAg, HBV DNA, or both)
7. HCV treatment or HCV RNA>LOD within the previous 6 months
8. Receipt of a licensed or Emergency Use Authorization vaccine within 4 weeks prior to study screening or plans to receive live attenuated vaccines within 4 weeks or any other licensed or Emergency Use Authorization vaccine within 2 weeks prior to or 2 weeks after any of the study investigational product administrations.
9. Plans to receive an MVA-vectored licensed or Emergency Use Authorization vaccine (i.e., smallpox or Mpox vaccine) within 12 weeks prior to or 2 weeks after either of the two study MVA.tHIVconsv4 vaccine administrations.
10. Receipt of an investigational study agent within 12 months prior to study screening Note: Receipt of a licensed vaccine as an investigational agent for an off-label indication is not exclusionary, subject to investigator discretion and the time limits in exclusion #8.
11. Previous receipt of immunoglobulin (IgG) therapy Note: Individuals who received IgGs as prophylactic therapy (e.g., for HBV or rabies exposure) >12 months prior to screening will not be excluded.
12. Previous receipt of humanized or human monoclonal antibody whether licensed or investigational Note: Individuals who received monoclonal antibody for the prevention and/or treatment of SARS-CoV-2/COVID-19 >12 months prior to screening will not be excluded.
13. Previous participation in a candidate HIV vaccine study or immune prophylaxis for HIV-1 infection with confirmed receipt of active product or with unknown receipt of active product vs placebo (i.e. remains blinded to what was actually received).
14. History of use of any immunomodulatory medications within 6 months of study entry including systemic corticosteroids (>14 days), immunosuppressants, anti-cancer drugs, interleukins, systemic interferons, systemic chemotherapy, or other medications that the site investigator feels could have an immune modulatory effect Note: Topical or inhaled corticosteroids are not prohibited.
15. Known allergy or history of anaphylaxis or other serious adverse reactions to vaccines, vaccine products, neomycin, streptomycin, gentamicin or egg products
16. History of a severe allergic reaction with generalized urticaria, angioedema or anaphylaxis in the 2 years prior to enrollment
17. History of chronic urticaria requiring daily treatment or a history of chronic or recurrent eczema and/or atopic dermatitis
18. History of splenectomy
19. Pregnant, breastfeeding or planning to become pregnant while enrolled in this study
20. Major psychiatric illness and/or substance use during the past 12 months that in the opinion of the investigator would preclude participation

Step 2 Inclusion Criteria (Group 3 only)

Group 3 will enter the study in Step 2. Participants are eligible to be included in the Group 3 protocol Step 2 only if all of the following criteria are met:

1. Thai National
2. Age ≥18 and ≤60 years of age
3. Can read and write Thai
4. Able and willing to provide written informed consent
5. The following laboratory values at screening:

   1. CD4 > 200 cells/mm3
   2. Absolute neutrophil count (ANC) ˃1,000/mm3
   3. Hemoglobin >11.5 g/dL
   4. Platelet count ˃150,000/mm3
   5. Estimated glomerular filtration rate (eGFR) ≥60 mL/min/1.73m2 using the re-expressed MDRD equation with Thai racial factor or the CKD-EPI Cystatin C equation
   6. Aspartate aminotransferase (AST) (SGOT), Alanine aminotransferase (ALT) (SGPT), alkaline phosphatase (AP), and total bilirubin <2x the upper limit of normal (ULN)
   7. HIV-1 RNA > 1,000 copies/mL
   8. HCV RNA negative
6. For persons of childbearing potential, negative pregnancy test at the screening visit.
7. Persons of childbearing potential must agree to not become pregnant and use two methods of contraception if engaging in sexual activity that could lead to pregnancy. Contraception must be used from the time of screening until the end of the study or until viral suppression in Step 4, whichever occurs first.
8. Participants engaging in sexual activity that could lead to pregnancy in the partner and who are of reproductive potential must agree to use a condom to avoid pregnancy in a spouse or partner of childbearing potential and to avoid transmitting HIV to an uninfected partner. A condom must be used from the time of screening until the end of the study or until viral suppression in Step 4, whichever occurs first.
9. Willingness to abstain from sexual intercourse, or use a condom, or partner(s) using pre-exposure prophylaxis consistently during ATI and until plasma HIV-1 RNA is less than limit of detection after ART restart with all partners that are HIV-uninfected or serostatus unknown.
10. Passes Test of Understanding (Protocol Section 8.4)
11. Willing to interrupt and restart ART according to study schedule
12. Willing to participate and adhere to the prohibitions and restrictions specified in this protocol for the duration of the study visits and follow up.
13. Experiencing early acute HIV-1 infection as defined by

    1. blood samples on at least two separate days positive by nucleic acid testing within 21 days of a negative nucleic acid HIV-1 test. OR
    2. by a positive nucleic acid test or a positive 4th generation EIA in the context of a negative 2nd or negative 3rd generation HIV-1 EIA test
14. No history of antiretroviral drug use for any indication in the last 30 days

Step 2 Exclusion Criteria (Group 3 only)

Participants who meet any of the following criteria will be excluded from the study for Group 3:

1. Weight <50 kg or > 115 kg
2. Presence of HLA B*57:01 allele associated with viral control.
3. Anyone with contraindication to intramuscular injections, placement of intravenous lines, and blood draws
4. Acute or serious illness requiring systemic treatment and/or hospitalization within 90 days prior to entry.
5. Any clinically significant acute or chronic medical condition, that in the opinion of the investigator would preclude participation including cardiovascular, pulmonary, hepatic, renal, gastrointestinal, genitourinary, hematological, coagulation, immunological disorders, that in the opinion of the investigator would preclude participation (e.g., history of seizure disorders, cardiovascular disease, bleeding/clotting disorder, autoimmune disease, malignancy, poorly controlled asthma, active tuberculosis or other systemic infections, etc.).
6. Active or chronic hepatitis B virus infection (detectable HBsAg)
7. HCV treatment or HCV RNA>LOD within the previous 6 months
8. Receipt of a licensed or Emergency Use Authorization vaccine within 4 weeks prior to study screening or plans to receive live attenuated vaccines within 4 weeks or any other licensed or Emergency Use Authorization vaccine within 2 weeks prior to or 2 weeks after any of the study investigational product administrations.
9. Plans to receive an MVA-vectored licensed or Emergency Use Authorization vaccine (i.e., smallpox or Mpox vaccine) within 12 weeks prior to or 2 weeks after either of the two study MVA.tHIVconsv4 vaccine administrations.
10. Receipt of an investigational study agent within 12 months prior to study screening Note: Receipt of a licensed vaccine as an investigational agent for an off-label indication is not exclusionary, subject to investigator discretion and the time limits in exclusion #8.
11. Previous receipt of immunoglobulin (IgG) therapy Note: Individuals who received IgGs as prophylactic therapy (i.e., for HBV or rabies exposure) >12 months prior to screening will not be excluded.
12. Previous receipt of humanized or human monoclonal antibody whether licensed or investigational Note: Individuals who received monoclonal antibody for the prevention and/or treatment of SARS-CoV-2/COVID-19 >12 months prior to screening will not be excluded.
13. Previous participation in a candidate HIV vaccine study or immune prophylaxis for HIV-1 infection with confirmed receipt of active product or with unknown receipt of active product vs placebo (i.e. remains blinded to what was actually received).
14. History of use of any immunomodulatory medications within 6 months of study entry including systemic corticosteroids (>14 days), immunosuppressants, anti-cancer drugs, interleukins, systemic interferons, systemic chemotherapy, or other medications that the site investigator feels could have an immune modulatory effect Note: Topical or inhaled corticosteroids are not prohibited.
15. Known allergy or history of anaphylaxis or other serious adverse reactions to vaccines, vaccine products, neomycin, streptomycin, gentamicin or egg products
16. History of a severe allergic reaction with generalized urticaria, angioedema or anaphylaxis in the 2 years prior to enrollment
17. History of chronic urticaria requiring daily treatment or a history of chronic or recurrent eczema and/or atopic dermatitis
18. History of splenectomy
19. Pregnant, breastfeeding or planning to become pregnant while enrolled in this study
20. Major psychiatric illness and/or substance use during the past 12 months that in the opinion of the investigator would preclude participation
21. Absolute neutrophil count (ANC) < 740 cells/mm3
22. Severe Acute Retroviral Syndrome requiring in-patient hospitalization or interfering with participant ability to return for follow-up visits.

Step 3 (ATI) Inclusion Criteria (All Groups) Step 3 will begin after the third and final vaccine (or placebo) administration (end of Step 2). Participant clinical status or laboratory tests may potentially change during Steps 1 and 2. To ensure that participants continue to meet safety criteria for proceeding to ATI, they will be screened (to include all required screening laboratory tests) for Step 3 inclusion criteria at the visit for the third and final vaccine/placebo dose (Last Step 2 visit): Step 2, Week 20 for Groups 1 and 2; Step 2, Week 28 for Group 3.

Participants enrolled in all Groups of the study may proceed with Step 3 if they meet all the following inclusion criteria:

1. Receipt of all doses of the study products and/or placebos per protocol in Steps 1 and 2.
2. Plasma HIV-1 RNA <50 copies/mL at the Last Step 2 visit.
3. CD4 T-cell count ≥400 cells/mm3 at the Last Step 2 visit. Note: The CD4 T-cell count can be repeated once, provided that the repeat is done within 4 weeks prior to Step 3 entry.
4. No CDC Category C event after study entry
5. Documented negative hepatitis B virus (HBV) surface antigen (HBsAg) at the Last Step 2 visit.
6. Documented negative hepatitis C virus (HCV) antibody (anti-HCV) or negative HCV RNA at the Last Step 2 visit.
7. For persons of childbearing potential, negative pregnancy test at the first Step 3 visit (Step 3, Week 0).
8. Persons of childbearing potential must agree to not become pregnant and use two methods of contraception if engaging in sexual activity that could lead to pregnancy.
9. Willingness to abstain from sexual intercourse, or use a condom, or partner(s) using pre-exposure prophylaxis consistently during ATI and until plasma HIV-1 RNA is less than limit of detection after ART restart with all partners that are HIV-uninfected or serostatus unknown.
10. Willingness to participate in ATI for up to 50 weeks.
11. Willingness to restart ART according to study guidelines.

Step 3 (ATI) Exclusion Criteria (All Groups)

Enrolled participants who meet any of the following criteria will be excluded from moving to Step 3:

1. Virologic failure (two consecutive HIV-1 RNA >1000 copies/mL) after study entry
2. Intercurrent illness, new medical diagnosis, laboratory abnormality, sign, or symptom that, in the opinion of the site investigator, would place participant at higher risk of morbidity during ATI.
3. Receipt of any non-nucleoside reverse transcriptase inhibitor (NNRTI) within 60 days before Step 3 entry.
4. Receipt of long-acting ART such as long-acting cabotegravir (CAB LA) or long-acting rilpivirine (RPV LA) at any point after study entry.
5. Failure by the participant to attend three consecutive Step 1 or Step 2 study visits.
6. Pregnancy or breastfeeding.
7. Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of VRC07-523LS and PGDM1400LS in combination with ChAdOx1.tHIVconsv1, ChAdOx1.HIVconsv62, MVA.tHIVconsv4 and A244d11 gp120/ALFQ vaccination in PLWH who initiated ART during AHI. | Measured from enrollment to a minimum of 50 weeks to a maximum of 100 weeks per participant
  Occurrence of ≥ grade 3 AE or SAE that are possibly, probably, or definitely related to the IPs during the study
To evaluate the impact of VRC07-523LS and PGDM1400LS in combination with ChAdOx1.tHIVconsv1, ChAdOx1.HIVconsv62, MVA.tHIVconsv4 and A244d11 gp120/ALFQ vaccination on viral load setpoint after viral rebound during ATI. | Measured for 50 weeks from entry into step 3 (treatment interruption and last mAb administration)
  Viral Load setpoint after 2 weeks post viral rebound during ATI.

SECONDARY OUTCOMES:
To evaluate the impact of VRC07-523LS and PGDM1400LS in combination with ChAdOx1.tHIVconsv1, ChAdOx1.HIVconsv62, MVA.tHIVconsv4 and A244d11 gp120/ALFQ vaccination on time to first documented HIV-1 RNA viral rebound of ≥50 copies/mL following ATI. | Measured for 50 weeks from entry into step 3 (treatment interruption and last mAb administration)
  Time (days) from ATI to first documented HIV-1 RNA viral rebound of ≥50 copies/mL
To evaluate the impact of VRC07-523LS and PGDM1400LS in combination with ChAdOx1.tHIVconsv1, ChAdOx1.HIVconsv62, MVA.tHIVconsv4 and A244d11 gp120/ALFQ vaccination on time to first documented HIV-1 RNA viral rebound of ≥1000 copies/mL following ATI. | Measured for 50 weeks from entry into step 3 (treatment interruption and last mAb administration)
  Time (days) from ATI to first documented HIV-1 RNA viral rebound of ≥1000 copies/mL
To evaluate the impact of VRC07-523LS and PGDM1400LS in combination with ChAdOx1.tHIVconsv1, ChAdOx1.HIVconsv62, MVA.tHIVconsv4 and A244d11 gp120/ALFQ vaccination on viral rebound dynamics during ATI. | Measured for 50 weeks from entry into step 3 (treatment interruption and last mAb administration)
  Peak viral load, nadir viral load, and viral load area under the curve (AUC) during the first 8 weeks after viral rebound.
To evaluate the impact of VRC07-523LS and PGDM1400LS in combination with ChAdOx1.tHIVconsv1, ChAdOx1.HIVconsv62, MVA.tHIVconsv4 and A244d11 gp120/ALFQ vaccination on the number of participants with plasma HIV-1 RNA < 1000 copies/mL at 12 and 24 weeks of | Measured for 50 weeks from entry into step 3 (treatment interruption and last mAb administration)
  The number of participants with plasma HIV-1 RNA < 1000 copies/mL at 12 and 24 weeks of ATI.
To evaluate the impact of VRC07-523LS and PGDM1400LS in combination with ChAdOx1.tHIVconsv1, ChAdOx1.HIVconsv62, MVA.tHIVconsv4 and A244d11 gp120/ALFQ vaccination on time to ART resumption for an HIV-related (virologic, immunologic, or clinical) reason d | i. Measured for 50 weeks from entry into step 3 (treatment interruption and last mAb administration)
  Time (days) from ATI to ART resumption during Step 3
To measure the effects of VRC07-523LS and PGDM1400LS in combination with ChAdOx1.tHIVconsv1, ChAdOx1.HIVconsv62, MVA.tHIVconsv4 and A244d11 gp120/ALFQ vaccination on HIV-1 RNA levels while on ART. | Measured for 50 weeks from entry into step 3 (treatment interruption and last mAb administration)
  HIV-1 RNA levels using single copy assay while on ART
To assess the impact of VRC07-523LS and PGDM1400LS in combination with ChAdOx1.tHIVconsv1, ChAdOx1.HIVconsv62, MVA.tHIVconsv4 and A244d11 gp120/ALFQ vaccination on total HIV-1 DNA levels prior to ATI | Measured for 50 weeks from entry into step 3 (treatment interruption and last mAb administration)
  Total HIV-1 DNA levels prior to ATI.
To assess the effects of VRC07-523LS and PGDM1400LS in combination with ChAdOx1.tHIVconsv1, ChAdOx1.HIVconsv62, MVA.tHIVconsv4 and A244d11 gp120/ALFQ vaccination on HIV-1 specific cellular immune responses prior to ATI. | Measure during step 2: from the initial administration of bNab therapy through week 22 in arms 1 and 2 and through week 30 in arm 3.
  Magnitude, breadth, cytokine production, cytotoxicity, proliferation and related functions of HIV-1 specific CD4 and CD8 T-cells prior to ATI.
To assess the effects of VRC07-523LS andPGDM1400LSin combination withChAdOx1.tHIVconsv1, ChAdOx1.HIVconsv62,MVA.tHIVconsv4 and A244d11 gp120/ALFQvaccination on HIV-1 specific humoral immuneresponses. | Measure at week 0 of Step 3 in all groups, just prior to ATI.
  Binding antibodies to HIV-1, ADCC, ADCP andother functional ab-mediated responses prior toATI.
To assess the impact of VRC07-523LS andPGDM1400LS in combination withChAdOx1.tHIVconsv1, ChAdOx1.HIVconsv62,MVA.tHIVconsv4 and A244d11 gp120/ALFQvaccination on the HIV-1 reservoir prior to ATI | Measure at week 0 of Step 3 in all groups, just prior to ATI.
  Measurements of HIV-1 reservoir using assaysbased on contemporary literature that may includebut are not limited to total and/or intact HIV-1DNA, quantitative infectious virus outgrowth(qVOA), cell- associated HIV-1 RNA, and relatedassays prior to ATI.
To characterize the pharmacokinetics of VRC07-523LS and PGDM1400LS. | Measure at week 0 of Step 3 in all groups, just prior to ATI.
  Levels of VRC07-523LS and PGDM1400LS
To describe the neurological, neuroimaging andneuro-cognitive effects that occur after receiptof VRC07-523LS and PGDM1400LS incombination with ChAdOx1.tHIVconsv1,ChAdOx1.HIVconsv62, MVA.tHIVconsv4 andA244d11 gp120/ALFQ vaccination and ATI | Measure at week 0 of Step 3 in all groups, just prior to ATI.
  Findings on CSF examination, MRI/MRS,neurological and neurocognitive testing before andafter receipt of study products and ATI
To assess the effects of VRC07-523LS and PGDM1400LSin combination with ChAdOx1.tHIVconsv1, ChAdOx1.HIVconsv62, MVA.tHIVconsv4 and A244d11 gp120/ALFQ vaccination on HIV-1 specific humoral immune responses. | Measure at week 0 of Step 3 in all groups, just prior to ATI.
  Measure Antibody Dependent Cellular Phagocytosis using clade AE protein coated target cells
To assess the impact of VRC07-523LS and PGDM1400LS in combination with ChAdOx1.tHIVconsv1, ChAdOx1.HIVconsv62, MVA.tHIVconsv4 and A244d11 gp120/ALFQ vaccination on the HIV-1 reservoir prior to ATI | Measure at week 0 of Step 3 in all groups, just prior to ATI.
  Total HIV intact DNA measured by the Intact Proviral DNA Assay
To assess the impact of VRC07-523LS and PGDM1400LS in combination with ChAdOx1.tHIVconsv1, ChAdOx1.HIVconsv62, MVA.tHIVconsv4 and A244d11 gp120/ALFQ vaccination on the HIV-1 reservoir prior to ATI | Measure at week 0 of Step 3 in all groups, just prior to ATI.
  Total HIV cell associate RNA measured by the quantitative RNA PCR
To characterize the pharmacokinetics of VRC07-523LS and PGDM1400LS. | Measured for 50 weeks from entry into step 3 (treatment interruption and last mAb administration)
  Concentration of PGDM1400LS during ATI by MSD

OTHER OUTCOMES:
To assess the impact of VRC07-523LS andPGDM1400LS in combination withChAdOx1.tHIVconsv1, ChAdOx1.HIVconsv62,MVA.tHIVconsv4 and A244d11 gp120/ALFQvaccination on the HIV reservoir when started at thetime of AHI and ART initiation | Measure at week 0 of Step 3 in all groups, just prior to ATI.
  Measurements of HIV-1 reservoir using assaysbased on contemporary literature that may includebut are not limited to total and/or intact HIV-1DNA, quantitative infectious virus outgrowth(qVOA), cell- associated HIV-1 RNA, and relatedassays prior to and following ATI
To assess the development of anti- drug antibody toVRC07-523LS and PGDM1400LS. | Measure at week 0 of Step 3 in all groups, just prior to ATI.
  Levels of ADA to VRC07-523LS andPGDM1400LS.
To evaluate baseline ChAdOx1 and ModifiedVaccinia Ankara (MVA) serostatus and its effects onimmune response and primary outcomes. | Measure at week 0 of Step 3 in all groups, just prior to ATI.
  ChAdOx1 nAbs titer at baseline and Vaccinia-virus-specific nAbs titer at baseline.
To characterize participant experiences in the trialand preferences about participation in HIV remissiontrials with treatment interruptions | Measured for 50 weeks from entry into step 3 (treatment interruption and last mAb administration)
  Responses to study participation questionnaires and pilot discrete choice experiment survey

CONTACTS AND LOCATIONS:
Locations (1):
- The Faculty of Medicine, Chulalongkorn University/ King Chulalongkorn Memorial Hospital, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No